CLINICAL TRIAL: NCT05412407
Title: What Are the Terms of Use of Analgesics for Acute Pain on a Patient Before a Consultation With a General Practitioner: Descriptive Epidemiological Study of Patients in General Practice in Rhône-Alpes
Brief Title: Analgesic Self-medication for Acute Pain by Patients Awaiting a Consultation With a General Practitioner
Acronym: AAPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0050
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain
Keywords: acute pain; analgesics; self medication
MeSH Terms: conditions — Acute Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire : Taken analgesics (Other): the patient will complete a questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — description of analgesic self-medication in the context of acute pain using a questionnaire evaluating the drug taken, the dosage, the duration of treatment, the type of pain, its intensity, the origin of the drug, the source of information consulted and the factors that prompted the patient to self-medicate

SUMMARY:
What are the terms of use of analgesics for acute pain on an outpatient basis before a consultation with a general practitioner? Descriptive epidemiological study of patients in general practice in Rhône-Alpes

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* without cognitive impairment
* having acute pain for less than 3 months
* Consultant to the practices participating to the study.

Exclusion Criteria:

* Patients who do not understand French
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-18 (Estimated); Primary Completion 2024-02-18 (Estimated); Study Completion 2024-02-18 (Estimated)

PRIMARY OUTCOMES:
Description of analgesic self-medication practices while waiting for a consultation with the general practitioner. | Inclusion
  dose of analgesic drugs per intake and per frequency

SECONDARY OUTCOMES:
Highlighting the reason for misuse of analgesics on an outpatient basis in the population studied while waiting for a consultation. | Inclusion
  Incidence of.each reason for misuse as indicated in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Assad ACHIQ, Principal Investigator — Médecins remplaçants
Locations (3):
- France (3):
  - MSP Hauteville, Hauteville-Lompnes
  - MSPU bel-air, Saint-Priest
  - Maison de santé de Malissol, Vienne

IPD SHARING:
Plan to Share IPD: No